CLINICAL TRIAL: NCT05977829
Title: Ultrasonographic, Hysteroscopic, Histopathologic Findings and Risk of Endometrial
Brief Title: Endometrial Malignancy in Breast Cancer Patients With or Without AUB
Acronym: TamAUB
Status: Completed | Type: Observational
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Gaetano Riemma, Principal Investigator, University of Campania Luigi Vanvitelli
Other Study IDs: 691
Record Dates: First submitted 2023-07-28; First posted 2023-08-04 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Endometrial Neoplasms
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Ultrasonography; Hysteroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Endometrial biopsy for histopathological analysis.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Breast cancer patients with abnormal uterine bleeding: * Transvaginal ultrasonography
  * Outpatient Hysteroscopy
  Interventions: Diagnostic Test: Ultrasound; Diagnostic Test: Hysteroscopy
- Breast cancer patients without abnormal uterine bleeding: * Transvaginal ultrasonography
  * Outpatient Hysteroscopy
  Interventions: Diagnostic Test: Ultrasound; Diagnostic Test: Hysteroscopy

INTERVENTIONS:
Diagnostic Test: Ultrasound — Transvaginal ultrasound to carry out uterine surveillance
Diagnostic Test: Hysteroscopy — Outpatient hysteroscopy to carry out uterine surveillance

SUMMARY:
In order to assess the hysteroscopic, histopathologic, and ultrasonographic aspects of uterine monitoring in postmenopausal breast cancer patients with or without abnormal uterine bleeding (AUB), as well as to calculate the risk of endometrial cancer in women with or without AUB.

DETAILED DESCRIPTION:
20-25% of postmenopausal women undergoing tamoxifen (TAM) therapy develop polyps, according to recent studies. Many large (>2 cm) and molecularly changed uterine polyps are usually seen in these women. Furthermore, a number of studies have demonstrated that TAM therapy raises the risk of endometrial cancer in both premenopausal and postmenopausal women. Studies suggest that women who use TAM may also have an increase in the prevalence of uterine sarcomas. In addition, the duration of TAM administration appears to increase the risk of endometrial cancer and uterine sarcoma.

This multicentric cohort study will compare the ultrasonographic, hysteroscopic, and histopathologic findings in postmenopausal women treated for breast cancer with or without AUB in order to increase the robustness of a still ambiguous literature on the subject. It will estimate the risk of endometrial cancer in women with AUB according to various covariates related to the breast neoplasm or the ultrasonographic and hysteroscopic features.

ELIGIBILITY:
Inclusion Criteria:

* In case of AUB: ultrasonographic endometrial thickness >5 mm at transvaginal ultrasound
* In case of non-AUB group ultrasonographic suspicion of endometrial or myometrial abnormalities

Exclusion Criteria:

* severe comorbidities (cardiovascular, metabolic, endocrine, and immunological disorders)
* receiving any other form of pharmacologic therapy

Ages: 43 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women undergoing gynecological examinations for endometrial surveillance related to selective estrogen receptor modulators, aromatase inhibitors or other hormone therapy for breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 283 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Endometrial cancer rate | 1 month after admission
Endometrial hyperplasia rate | 1 month after admission

CONTACTS AND LOCATIONS:
Overall Officials: Gaetano Riemma, MD, Principal Investigator — University of Campania Luigi Vanvitelli; Pasquale De Franciscis, MD PhD, Study Chair — University of Campania Luigi Vanvitelli
Locations (1):
- University of Cagliari, Cagliari, Italy